CLINICAL TRIAL: NCT05545839
Title: TRACER: Transition to Adulthood Through Coaching and Empowerment in Rheumatology, A Feasibility Study
Brief Title: Transition to Adulthood Through Coaching and Empowerment in Rheumatology
Acronym: TRACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Western University (Other)
Responsible Party: Principal Investigator, Michelle Batthish, Associate Professor, McMaster University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14499
Record Dates: First submitted 2022-09-13; First posted 2022-09-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Juvenile Idiopathic Arthritis; Juvenile Rheumatoid Arthritis; Juvenile Dermatomyositis; Juvenile Psoriatic Arthritis; Autoinflammatory Disease; Autoimmune Diseases; Lupus Erythematosus
Keywords: transition care; transition coaching
MeSH Terms: conditions — Arthritis, Juvenile; Dermatomyositis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care - control (No Intervention): Standard of care, appointments with adult rheumatology
- Transition coaching - experimental (Experimental): Participants will receive 8 transition coaching sessions (1/month) in addition to standard care
  Interventions: Behavioral: Transition coaching

INTERVENTIONS:
Behavioral: Transition coaching — Transition coaching sessions (8 sessions), covering paediatric to adult care, self-advocacy, medication management, general health, lifestyle and behaviours, future planning, screening for mood disorders and coping skills.
  Arms: Transition coaching - experimental

SUMMARY:
TRACER is a study aiming to investigate the feasibility of transition coaching sessions for patients moving from paediatric to adult rheumatology care.

DETAILED DESCRIPTION:
TRACER is a feasibility study investigating transition coaching for patients with rheumatic disease transferring from paediatric to adult rheumatology care. This is a vulnerable time in the patients' care and life as they are assuming more responsibility for their health and undergoing significant life transitions. There is risk for increased morbidity and mortality around this time if the patient are not well supported and if they do not stay engaged with care. This intervention aim to provide self-efficacy, self-management, coping skills and support to patients making the transition. This study aims to assess the feasibility of conducting a multi-centre randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pediatic-onset rheumatic disease
* At their last paediatric rheumatology appointment prior to transferring to adult rheumatology care
* Able to communicate in English
* Have a phone or device capable of participating in video conference
* Available over the next 8 months

Exclusion Criteria:

* Cognitive impairment preventing participation in individualized education sessions (as determined by medical staff)

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Consent rate | 19 month recruitment period
  % of patients approached who consent to the study
Enrolment from non-primary site | 19 month
  % of patients enrolled from non-primary site
Virtual session attendance | 3 year study period
  % of transition coaching sessions attended
Outcome measure completion | 3 year study period
  % of outcome assessments completed at 8 months (end of transition coach invention)
Missing data | 3 year study period
  % of missing data

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire | 3 year study period
  Descriptive statistics of PROMIS questionnaire (person-centered measures to assess how people feel and function) results at baseline, 8 months and 11 months, between the two groups.
Physician Global Assessment (PGA) | 3 year study period
  Descriptive statistics of physical global assessment at baseline and at subsequent follow-up, between the two groups. Physician Global Assessment refers to MD assessment of disease activity and is rated between 0 (no disease activity) and 10 (most active disease).
Active joint count | 3 year study period
  Descriptive statistics of active joint count (joints with evidence of active inflammation - including swelling, tenderness, loss of ROM) at baseline and at subsequent follow-up, between the two groups
Global function/quality of life | 3 year study period
  Descriptive statistics of PedsQL (Paediatric Quality of Life Inventory) 4.0 Generic Core Scales Young Adult Version questionnaire results at baseline, 8 months and 11 months, between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Batthish, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital at London Health Sciences Centre, London, Ontario